CLINICAL TRIAL: NCT00549627
Title: Evaluation of the PediGuard™ for Pedicle Screw Insertion
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: New funding sources being sought
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Randal Betz, MD, Shriners Hospitals for Children
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 4727
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Posterior Spinal Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pediguard — PediGuard™ is a hand-held drilling tool that allows real-time detection of vertebral pedicle and body breaches in all directions.

SUMMARY:
The aim of the study is to determine the relative effectiveness of the PediGuardTM , a device manufactured by SpineVision, Inc, for placement of a pedicle screw pilot (drill) hole and for reducing pedicle screw breaches during thoracic and lumbar pedicle screw fixation of the spine.

Hypothesis #1 The PediGuardTM will be more accurate for pedicle screw placement as compared to other standard manual techniques of similar size of pedicle screw insertion. At least 90% of screws placed with the PediGuardTM will be positioned correctly in the pedicle (defined as less than 2 mm breach by CT scan). In contrast, only 80% of screws using manual placement will be positioned correctly in the pedicle.

Hypothesis #2 The PediGuardTM will not be inferior to fluoroscopic techniques for pedicle screw insertion. Both techniques will achieve at least 90% accuracy in the placement of pedicle screws.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary spinal fusion with pedicle screw fixation of the spine anywhere from T1to S1
* Subjects must be skeletally mature as defined by closed growth plates on wrist via radiographs
* Written informed consent and assent (assent for adolescents)

Exclusion Criteria:

* Pedicle screw insertion by image guided techniques, including Fluoronav
* Tumor
* Diagnoses associated with diminished bone mineral density such as osteogenesis imperfecta, severe osteopenia, neurofibromatosis
* Severe senile osteoporosis (> 2 standard deviations below the norm)
* Women who are pregnant
* Children with open growth plates
* Previously fused spinal levels
* Unwillingness to sign written informed consent and assent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2005-08; Primary Completion 2008-11 (Actual); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
At least 90% of screws placed with the PediGuard™ will be positioned correctly in the pedicle (defined as less than 2 mm breach by CT scan). | Post-op CT prior to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Randal Betz, MD, Principal Investigator — Shriners Hospitals for Children
Locations (7):
- United States (6):
  - Panorama Orthopedics and Spine Center, Golden, Colorado
  - Miami Children's Hospital, Miami, Florida
  - University of Miami, Miami, Florida
  - Spine Institute, Louisville, Kentucky
  - NYU Hospital for Joint Diseases, New York, New York
  - Shriners Hospitals for Children, Philadelphia, Pennsylvania
- Victoria Hospital, London, Ontario, Canada